CLINICAL TRIAL: NCT02719821
Title: Refining a Biobehavioral Intervention to Enhance Recovery Following Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW15080; P30CA014520 (NIH); NCI-2016-00238 (Registry Identifier: CTRP); 2015-1261 (Other: IRB); 4UL1TR000427-10 (NIH); A538900 (Other: UW Madison); SMPH\PSYCHIATRY\PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-02

CONDITIONS: Hodgkin's Lymphoma; Leukemia; Lymphoid Leukemia; Multiple Myeloma; Myeloid Leukemia; Non-hodgkin's Lymphoma; Myelodysplastic Syndrome
Keywords: Hematopoietic Stem Cell Transplantation; Fatigue; Insomnia; Depression; Behavioral Intervention
MeSH Terms: conditions — Hodgkin Disease; Leukemia; Leukemia, Lymphoid; Multiple Myeloma; Leukemia, Myeloid; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Fatigue; Sleep Initiation and Maintenance Disorders; Depression | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Individuals treated with HSCT will learn behavioral techniques to improve sleep and increase daytime activity with the goal of alleviating insomnia, fatigue, and depression. Study investigators will conduct semi-structured interviews after each session to determine participant satisfaction with and acceptability of the behavioral strategies, timing, delivery mode, assessment strategy, and time commitment. Participants will be asked to complete a daily checklist indicating which intervention strategies they used daily. Participants will be asked to complete self-report assessments, to wear a wrist-worn actigraphy device, and to complete a sleep log at three time points: prior to HSCT and approximately 9 and 18 weeks post-HSCT.
  Interventions: Behavioral: Behavioral techniques

INTERVENTIONS:
Behavioral: Behavioral techniques — Learning behavioral techniques designed to improve nighttime sleep quality and daytime activity for approximately 45-60 minutes on three occasions.
  Device: Actiwatch-2 (Philips Respironics)

SUMMARY:
The goal of this project is to refine and evaluate the feasibility of a brief, behavioral intervention to improve the recovery following hematopoietic stem cell transplantation (HSCT). Cancer patients who were treated with HSCT will learn behavioral techniques to improve sleep and increase daytime activity with the goal of alleviating insomnia, fatigue, and depression after HSCT. If the intervention is feasible and acceptable to patients, a future study will test the effects in a larger trial, with the long-term goal of improving the care and quality of life of cancer survivors recovering from HSCT.

DETAILED DESCRIPTION:
Details of the assessment strategy:

Patient-reported outcomes:

Participants will complete self-report measures prior to HSCT and 9 (mid-intervention) and 18 weeks (post-intervention) post-HSCT. The sleep disturbance, fatigue, and depression modules of the NIH Patient Reported Outcomes Measurement Information System (PROMIS) will be the primary outcomes. The investigators will compare performance with more established instruments the investigation team has previously used: Insomnia Severity Index (ISI), Fatigue Symptom Inventory (FSI), and the Inventory of Depression and Anxiety Symptoms (IDAS) depression subscale.

Actigraphy:

The Actiwatch-2 (Philips Respironics), a wrist-worn actigraphy device, will be used to objectively quantify circadian rest-activity patterns over a continuous 7-day period using 1-minute sampling epochs at three time points: prior to HSCT and 9 (mid-intervention) and 18 weeks (post-intervention) post-HSCT. The following indices will be calculated: mesor (mean activity level), amplitude (rhythm height), acrophase (time of day the rhythm peaks), and R-squared (robustness of the rhythm). Participants will complete a concurrent nightly sleep log, and traditional sleep parameters will be calculated from both the logs and actigraphy, including total sleep time (TST), sleep onset latency (SOL), wake time after sleep onset (WASO), and sleep efficiency (SE). For daytime activity, calibration thresholds will be used to aggregate activity data into steps and minutes spent in sedentary, light, moderate, and vigorous activity

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older undergoing hematopoietic stem cell transplantation (HSCT) at the University of Wisconsin Carbone Cancer Center (UWCCC)
* Autologous transplant recipients with multiple myeloma or lymphoma (both Hodgkin's and Non-Hodgkin's types) receiving standard conditioning regimens
* Allogeneic transplant recipients undergoing fully ablative transplants
* Participants who develop treatment complications or disease recurrence after being enrolled in the study may continue to participate if they are able to do so

Exclusion Criteria:

* Autologous transplant recipients receiving non-standard regimens
* Autologous transplant recipients with diagnoses other than multiple myeloma or lymphoma
* Allogeneic transplant recipients receiving reduced intensity regimens

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Ability to recruit, retain, and collect complete data from all participants | 18 weeks
  Recruitment rate, reasons for non-participation, and attrition will be tracked at Retention rates and those contributing complete data will be tracked at milestones throughout the study period.
Intervention uptake and adherence | 18 weeks
  Participants will be asked to complete a daily checklist to indicate which intervention strategies they attempted each day.
Intervention fidelity | 18 weeks
  A selection of audio recorded intervention sessions will be evaluated using a fidelity checklist.
Participant satisfaction and acceptability | 18 weeks
  Study investigators will conduct semi-structured interviews approximately one week after each session to determine participant satisfaction with and acceptability of the behavioral strategies, timing, delivery mode, assessment strategy, and time commitment; the interviews will be audio recorded. Participants will be asked about barriers to participation and problems encountered as well as areas of satisfaction with each of the aforementioned elements. Recordings will be reviewed to generate a list of barriers and facilitators of participation.
Acceptability of the assessment strategy | 18 weeks
  Acceptability will be assessed by examining the aforementioned semi-structured interview data and rates of completion of self-report measures and actigraphy.
  We will examine rates of completion of the following self-report measures:
  NIH Patient Reported Outcomes Measurement Information System (PROMIS) sleep disturbance, fatigue, and depression modules; Insomnia Severity Index (ISI); Fatigue Symptom Inventory (FSI); Inventory of Depression and Anxiety Symptoms (IDAS) depression subscale
  We will examine rates of completion of sufficient actigraphy data for calculating the following indices:
  Mesor (mean activity level); Amplitude (rhythm height); Acrophase (time of day the rhythm peaks); R-squared (robustness of the rhythm); total sleep time (TST); sleep onset latency (SOL); wake time after sleep onset (WASO); sleep efficiency (SE)
Validity of the assessment strategy | 18 weeks
  To address validity, the investigators will assess the ability of PROMIS measures to predict legacy measures the investigators have previously used successfully with this patient population (ISI, FSI, IDAS).

CONTACTS AND LOCATIONS:
Overall Officials: Erin Costanzo, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252